CLINICAL TRIAL: NCT01615939
Title: A Randomized Controlled Trial Comparing Continuous Sciatic Nerve Block to Single Shot Sciatic Nerve Block
Brief Title: A Study Comparing Continuous Sciatic Nerve Block to Single Shot Sciatic Nerve Block
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study has been terminiated due to minimal subject recruitment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Antoun Nader, Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00058306; STU00058306
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Results first posted 2016-06-30 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-06

CONDITIONS: Fracture of Foot
Keywords: Sciatic Nerve Block; Continuous Nerve Block
MeSH Terms: interventions — Bupivacaine; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Shot Sciatic Nerve Block (Active Comparator): Single shot sciatic nerve blocks will be performed by resident trainees supervised by faculty. Bupivacaine 0.625% with epinephrine 1:300,000 will be injected incrementally in 3-ml aliquots to a total volume of 0.4 ml/kg (minimum, 20 ml; maximum, 35 ml).
  Interventions: Drug: Bupivacaine
- Continuous Sciatic Nerve Block (Active Comparator): Continuous sciatic nerve block catheters will be performed using an insulated needle connected to the negative lead of a constant current nerve stimulator. The catheter will be advanced under ultrasound guidance. A test dose of 1.5% lidocaine with epinephrine will be injected to confirm catheter placement. All subjects will receive a portable pump that will infuse 0.2% ropivacaine 5 ml/hr with a 5 ml bolus/hr. The subjects will follow standard protocol discharge instructions in regards to removing the catheter themselves.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine 0.625% with epinephrine 1:300,000
  Other Names: Sensorcaine
  Arms: Single Shot Sciatic Nerve Block
Drug: Ropivacaine — 0.2% ropivacaine 5 ml/hr with a 5 ml bolus/hr.
  Other Names: Naropin
  Arms: Continuous Sciatic Nerve Block

SUMMARY:
The purpose of this study is to compare the incidence of postoperative symptoms of neurologic injury after a single shot infragluteal-parabiceps sciatic nerve block versus a continuous infragluteal-parabiceps sciatic nerve catheter.

DETAILED DESCRIPTION:
There are a limited number of prospective studies in the literature examining the risk of neurologic injury and symptoms after sciatic nerve blocks. The incidence of transient neurological symptoms after a continuous catheter is not well reported.

ELIGIBILITY:
Inclusion Criteria:

* all patients ( ≥18 and ≤ 80) who are scheduled to undergo elective scheduled foot surgery and agreed to receive a sciatic nerve catheter as a part of their postoperative pain management. this study.

Exclusion Criteria:

* history of hemostatic abnormalities
* chronic pain syndrome
* a foot deformity restricting normal foot movement
* severe liver or renal disease
* a preexisting neurologic disorder
* patient refusal to participate
* the presence of language barrier that prohibits proper communication with patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoun Nader, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Shot Sciatic Nerve Block | Continuous Sciatic Nerve Block
Started | 13 | 4
Completed | 8 | 4
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Shot Sciatic Nerve Block | Continuous Sciatic Nerve Block | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 3 | 1 | 4
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [33 to 73] | 41 [30 to 61] | 41 [33 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Temporary Neurologic Symptoms Between Groups
Description: Temporary neurologic symptoms between groups; muscle weakness of either foot dorsiflexion and plantar flexion
Time Frame: 1 month
Measure: Number; unit: percentage of total participants
Arm/Group | Single Shot Sciatic Nerve Block | Continuous Sciatic Nerve Block
Number analyzed (Participants) | 8 | 4
percentage of total participants | 0 | 0

2. Secondary Outcome: Participant Satisfaction With Anesthesia
Description: Patient satisfaction on a 0 to 10 scale with 0 equals completely dissatisfied and 10 equals completely satisfied
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Single Shot Sciatic Nerve Block | Continuous Sciatic Nerve Block
Number analyzed (Participants) | 8 | 4
units on a scale | 10 [10 to 10] | 10 [10 to 10]

3. Secondary Outcome: Pain Control
Description: Numeric rating score for pain (NRS) 0 to 10 scale where 0 equals no pain and 10 equals the worst pain imaginable
Time Frame: 72 hrs
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Single Shot Sciatic Nerve Block | Continuous Sciatic Nerve Block
Number analyzed (Participants) | 8 | 4
units on a scale | 5 [1 to 6] | 6 [3 to 8]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Single Shot Sciatic Nerve Block | Continuous Sciatic Nerve Block
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 0/4

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes